CLINICAL TRIAL: NCT00906555
Title: The Effect of Different Dosages of Solute Clearance on Outcome in Twice Weekly Hemodialysis Patients-A Prospective, Randomized, Multi-center Intervention Study
Brief Title: The Effect of Different Dosages of Solute Clearance on Outcome in Twice Weekly Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Aiwu Lin, Vice Director, Department of Nephrology, Renji Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08dz1900501-a
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Renal Replacement Therapy; Hemodialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): hemodialysis patients with baseline Kt/V between 1.2 and 1.7 (1.2 ≤ Kt/V < 1.7)
- 2 (Experimental): Modification of hemodialysis parameters such as dialysis time, blood flow rate and dialysate flow rate to reach a Kt/V ≥ 1.7.
  Interventions: Procedure: modification of hemodialysis parameters on dialysis machine

INTERVENTIONS:
Procedure: modification of hemodialysis parameters on dialysis machine — Modification of hemodialysis parameters such as dialysis time, blood flow rate and dialysate flow rate to reach a Kt/V ≥ 1.7.
  Arms: 2

SUMMARY:
Adequacy of solute clearance makes a profound impact on clinical outcome in maintenance hemodialysis patients. Thus far, guidelines on the target of solute clearance (Kt/V or URR) are based on patients with three dialysis sessions per week. However, quite a few patients have their dialysis sessions twice per week in China. The dialysis target of solute clearance in this population remains to be elucidated. The aim of this study was to explore the optimum target solute clearance (Kt/V or URR) in maintenance hemodialysis patients with two dialysis sessions per week. Two groups of hemodialysis patients with different Kt/V (1.2 ≤ Kt/V < 1.7 versus Kt/V ≥ 1.7) will be followed until 96 weeks in this prospective, randomized, multi-center, interventional study.

DETAILED DESCRIPTION:
This is a prospective, randomized, multi-center intervention study. 400 maintenance hemodialysis patients with twice dialysis sessions per week will be enrolled into the study. All the patients have their baseline Kt/V between 1.2 and 1.7 (1.2 ≤ Kt/V < 1.7). After treatment intervention, the patients will be randomized to two groups according to their different Kt/V (1.2 ≤ Kt/V < 1.7 vs. Kt/V ≥ 1.7), then the patients will be regularly followed up at baseline, 12 weeks, 24 weeks, 48 weeks, 72 weeks and 96 weeks. Clinical outcomes such as mortality, complications and life quality between the two groups will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing maintenance hemodialysis for more than 12 weeks were included in the study.
2. The patients have their dialysis sessions twice weekly and have baseline Kt/V between 1.2 and 1.7 (1.2 ≤ Kt/V < 1.7).
3. Age from 18 to 80, male or female.
4. Patients have long term vascular access.

Exclusion Criteria:

1. Patients with an expected survival less than 12 months.
2. Without informed consent.
3. Unstable organ disease such as uncurable cancer,active inflammation disease and mental disease.
4. Patients with an expected follow up less than 48 weeks,such as planned kidney transplant.
5. Other conditions regarded as unsuitability by investigator, such as pregnancy, alcohol or drug indulgence. A dry weight more than 90 kg is also excluded in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2009-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
clinical outcome including mortality and morbidity | 2 years

SECONDARY OUTCOMES:
complications including cardiovascular disease, nutritional and inflammation status, calcium and phosphorus level, anemia and life quality | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jiaqi Qian, MD, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University school of medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No